CLINICAL TRIAL: NCT00441233
Title: Clinical Performance of Extended Wear Silicone Hydrogel Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: Menicon Co., Ltd. (Industry); Clinical Vision Research Australia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H07 001
Record Dates: First submitted 2007-02-27; First posted 2007-02-28 (Estimated); Last update posted 2008-01-09 (Estimated); Status verified 2007-12

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

INTERVENTIONS:
Device: Silicone hydrogel contact lens

SUMMARY:
The primary purpose of this study is to investigate the clinical performance of a new silicone hydrogel contact lens over a period of 6 months of extended wear.

ELIGIBILITY:
Inclusion Criteria:

* Is correctable to at least 6/9 distance visual acuity in each eye with spherical contact lenses.
* Is a current daily wear soft contact lens wearer.
* Has no clinically significant anterior eye findings.
* Has no other active ocular disease.

Exclusion Criteria:

* Has any systemic disease that might interfere with contact lens wear
* Is using any systemic or topical medications that will affect ocular health.
* Has any pre-existing ocular irritation that would preclude contact lens fitting.
* Has any ocular pathology or severe insufficiency of lacrimal secretion (dry eyes) that would affect the wearing of contact lenses.
* Has undergone corneal refractive surgery.
* Is pregnant, lactating or planning a pregnancy.

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Dates: Start 2007-03; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Lakkis, BScOptom, PhD, PGCertOcTher, Principal Investigator — Clinical Vision Research Australia, University of Melbourne
Locations (1):
- Clinical Vision Research Australia, Melbourne, Victoria, Australia